CLINICAL TRIAL: NCT01855477
Title: Development of a Platform for Next-generation DNA Sequencing Based Personalized Treatment for Cancer Patients: Protocol to Obtain Biopsies From Patients With Locally Advanced or Metastatic Cancer (CPCT - 02 Biopsy Protocol)
Brief Title: CPCT-02 Biopsy Protocol
Acronym: CPCT-02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation CPCT (Other)
Collaborators: Hartwig Medical Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL35781.041.11
Record Dates: First submitted 2013-05-13; First posted 2013-05-16 (Estimated); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Solid Tumors; Metastatic Disease
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Histological biopsy procedure (Other): This is a multicenter study combining histological biopsy of tumor material with DNA sequencing using Next Generation Sequencing (NGS) platform. The study aims to obtain a more accurate pre-treatment stratification of cancer patients by obtaining fresh tumor biopsies for next-generation sequencing to obtain a mutational profile.
  Interventions: Procedure: Histological biopsy procedure

INTERVENTIONS:
Procedure: Histological biopsy procedure

SUMMARY:
A major challenge for researchers in cancer care is to expedite the development of new therapeutics and the Center for Personalized Cancer Treatment (a collaboration of the Dept. of Medical Oncology from the University Medical Center Utrecht, Netherlands Cancer Center - Antoni van Leeuwenhoek hospital and the Erasmus Medical Center - Daniël den Hoed clinic) is an initiative to achieve this goal.

The current and future generation anti-cancer drugs are developed to specifically activate or deactivate deregulated gene products or signaling pathways in cancer cells. The development of such "targeted" agents is an exciting new opportunity that promises to deliver more anti-cancer efficacy and less toxicity. Although targeted therapy has been a breakthrough in medical oncology leading to the development of a portfolio of potentially successful new drugs, it has not yet delivered the much needed relief for large patient populations. We believe that the development of these agents is mainly hampered by our lack of successful patient selection.

The CPCT aims to select patients for clinical trial participation based on the results of Next Generation Sequencing (NGS) information obtained from tumor material. The advent of NGS platforms enables us to probe a significant proportion of the cancer genome and thus to develop a realistic view on the complex genetic changes in cancer cells. The CPCT aims to use NGS platforms to improve the selection of patients for targeted therapy trials.

We will obtain tumor biopsies of a (preferably) metastatic or locally advanced lesion and peripheral blood sample from all patients included in the trial; the biopsies to obtain information on the tumor related genetic mutations (mutational profile) and the blood samples to assess each patient's germline DNA background variation. As patients will be asked to undergo an invasive procedure it is important to address the potential safety issues. Review of the literature shows that in general tumor biopsies can be performed with only minor complications and acceptable risks. We will recruit patients with metastatic or locally advanced (incurable) solid tumors and we aim to use the information obtained from DNA sequencing to stratify patients for inclusion in clinical trials. The final personalized treatment decision will be made dependent on the availability of trials and the expected predictive value of the mutational profile.

ELIGIBILITY:
Selection criteria, defined as inclusion criteria, are:

1. Patients with the following locally advanced or metastatic cancer for whom a new line of therapy is indicated below starting within 3 months after biopsy (see also table 2):

   - Metastatic Pancreas Cancer: FOLFIRINOX (Folinic acid [leucovorin] + Fluorouracil [5-FU] + Irinotecan + Oxaliplatin)
2. Measurable metastatic or locally advanced lesion(s), according to RECIST 1.1 criteria18. Guidelines for response evaluation are given in appendix A.
3. Metastatic or locally advanced lesion(s) of which a histological biopsy can safely be obtained.
4. Patients age > 18 years, willing and able to comply with the protocol as judged by the investigator with a signed informed consent.

Patients must meet selection criteria 3 not only prior to baseline biopsy, but also prior to the (optional and if applicable, see CPCT-02 Study manual) post-treatment biopsies.

Exclusion criteria:

* If one or more of the above mentioned inclusion criteria is not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6927 (Actual)
Dates: Start 2011-08-17 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
• Percentage of patients enrolled in clinical intervention trials based on the mutational profile of their cancer genome | 3 months after baseline biopsy

SECONDARY OUTCOMES:
Percentage of samples with sufficient DNA for sequencing analysis | 1 year after baseline biopsy
• Percentage of samples with an adequate mutational profile to allow enrollment in trials | 1 year after baseline biopsy
Differences in mutational profile pre, post and during treatment | 1 year after last biopsy within one line of treatment
• Number and nature of (serious) adverse events of the performed histological biopsies | 14 days after each biopsy procedure

CONTACTS AND LOCATIONS:
Overall Officials: Haiko HJ Bloemendal, Prof. Dr., Study Director — Radboud University Medical Center
Locations (1):
- Foundation CPCT, Radboud UMC, Nijmegen, South Holland, Netherlands

REFERENCES:
- [Derived] Vis DJ, Palit SAL, Corradi M, Cuppen E, Mehra N, Lolkema MP, Wessels LFA, van der Heijden MS, Zwart W, Bergman AM. Whole genome sequencing of 378 prostate cancer metastases reveals tissue selectivity for mismatch deficiency with potential therapeutic implications. Genome Med. 2025 Mar 20;17(1):24. doi: 10.1186/s13073-025-01445-5. PMID 40114169
- [Derived] van de Haar J, Mankor JM, Hummelink K, Monkhorst K, Smit EF, Wessels LFA, Cuppen E, Aerts JGJV, Voest EE. Combining Genomic Biomarkers to Guide Immunotherapy in Non-Small Cell Lung Cancer. Clin Cancer Res. 2024 Apr 1;30(7):1307-1318. doi: 10.1158/1078-0432.CCR-23-4027. PMID 38300729
- [Derived] Verschoor N, Smid M, Jager A, Sleijfer S, Wilting SM, Martens JWM. Integrative whole-genome and transcriptome analysis of HER2-amplified metastatic breast cancer. Breast Cancer Res. 2023 Nov 15;25(1):145. doi: 10.1186/s13058-023-01743-z. PMID 37968696
- [Derived] de Joode K, van de Geer WS, van Leenders GJLH, Hamberg P, Westgeest HM, Beeker A, Oosting SF, van Rooijen JM, Beerepoot LV, Labots M, Mathijssen RHJ, Lolkema MP, Cuppen E, Sleijfer S, van de Werken HJG, van der Veldt AAM. The genomic and transcriptomic landscape of advanced renal cell cancer for individualized treatment strategies. Sci Rep. 2023 Jul 3;13(1):10720. doi: 10.1038/s41598-023-37764-z. PMID 37400554
- [Derived] Nakauma-Gonzalez JA, Rijnders M, van Riet J, van der Heijden MS, Voortman J, Cuppen E, Mehra N, van Wilpe S, Oosting SF, Rijstenberg LL, Westgeest HM, Zwarthoff EC, de Wit R, van der Veldt AAM, van de Werken HJG, Lolkema MPJ, Boormans JL. Comprehensive Molecular Characterization Reveals Genomic and Transcriptomic Subtypes of Metastatic Urothelial Carcinoma. Eur Urol. 2022 Apr;81(4):331-336. doi: 10.1016/j.eururo.2022.01.026. Epub 2022 Jan 25. PMID 35086719
- [Derived] Roepman P, de Bruijn E, van Lieshout S, Schoenmaker L, Boelens MC, Dubbink HJ, Geurts-Giele WRR, Groenendijk FH, Huibers MMH, Kranendonk MEG, Roemer MGM, Samsom KG, Steehouwer M, de Leng WWJ, Hoischen A, Ylstra B, Monkhorst K, van der Hoeven JJM, Cuppen E. Clinical Validation of Whole Genome Sequencing for Cancer Diagnostics. J Mol Diagn. 2021 Jul;23(7):816-833. doi: 10.1016/j.jmoldx.2021.04.011. Epub 2021 May 6. PMID 33964451
- [Derived] Mendelaar PAJ, Smid M, van Riet J, Angus L, Labots M, Steeghs N, Hendriks MP, Cirkel GA, van Rooijen JM, Ten Tije AJ, Lolkema MP, Cuppen E, Sleijfer S, Martens JWM, Wilting SM. Whole genome sequencing of metastatic colorectal cancer reveals prior treatment effects and specific metastasis features. Nat Commun. 2021 Jan 25;12(1):574. doi: 10.1038/s41467-020-20887-6. PMID 33495476